CLINICAL TRIAL: NCT04075305
Title: The Multiple Outcome Evaluation of Radiation Therapy Using the MR-Linac Study
Brief Title: The MOMENTUM Study: The Multiple Outcome Evaluation of Radiation Therapy Using the MR-Linac Study
Acronym: MOMENTUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: The Netherlands Cancer Institute (Other); Sunnybrook Health Sciences Centre (Other); M.D. Anderson Cancer Center (Other); The Christie NHS Foundation Trust (Other); Royal Marsden NHS Foundation Trust (Other); Medical College of Wisconsin (Other); Elekta Limited (Industry); Odense University Hospital (Other); Radboud University Medical Center (Other); Radiotherapiegroep (Other); Jules Bordet Institute (Other); University Hospital Tuebingen (Other); Radiotherapeutic Institute Friesland (Other); Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other); IRCCS Sacro Cuore Don Calabria di Negrar (Other); Austin Health (Other Government); Princess Margaret Hospital, Canada (Other); Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, Helena M Verkooijen, Prof. Dr., UMC Utrecht
Other Study IDs: NL66650.041.18
Record Dates: First submitted 2019-03-22; First posted 2019-08-30 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Oncology; Breast Cancer; Prostate Cancer; Gynecologic Cancer; Brain Tumor; Brain Cancer; Gynecologic Tumor; Prostate Tumor; Prostate Neoplasm; Breast Tumor; Radiation Toxicity; Quality of Life; Rectal Cancer; Rectal Tumor; Rectal Neoplasms; Lung Cancer; Lung Tumor; Lung Neoplasm; Esophageal Cancer; Esophagus Cancer; Esophageal Tumor; Esophageal Neoplasm; Esophagus Tumor; Esophagus Neoplasm; Pancreatic Cancer; Pancreatic Tumor; Pancreatic Neoplasms; Head and Neck Cancer; Head and Neck Neoplasms; Head and Neck Tumor; Tumor; Neoplasms; Bladder Cancer; Bladder Neoplasm; Liver Cancer; Liver Neoplasms; Liver Metastases; Oligometastases
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Brain Neoplasms; Genital Neoplasms, Female; Radiation Injuries; Rectal Neoplasms; Lung Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Head and Neck Neoplasms; Urinary Bladder Neoplasms; Liver Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (13):
- Brain cancer
  Interventions: Radiation: Radiation therapy
- Lung cancer
  Interventions: Radiation: Radiation therapy
- Esophageal cancer
  Interventions: Radiation: Radiation therapy
- Breast Cancer
  Interventions: Radiation: Radiation therapy
- Head and Neck Cancer
  Interventions: Radiation: Radiation therapy
- Pancreatic cancer
  Interventions: Radiation: Radiation therapy
- Gynecological cancer
  Interventions: Radiation: Radiation therapy
- Rectal cancer
  Interventions: Radiation: Radiation therapy
- Prostate cancer
  Interventions: Radiation: Radiation therapy
- Bladder cancer
  Interventions: Radiation: Radiation therapy
- Oligometastases
  Interventions: Radiation: Radiation therapy
- Liver cancer
  Interventions: Radiation: Radiation therapy
- Other types of cancer
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy on the CE marked and FDA approved MR-Linac

SUMMARY:
The Multi-OutcoMe EvaluatioN of radiation Therapy Using the Unity MR-Linac Study (MOMENTUM) is a multi-institutional, international registry facilitating evidenced based implementation of the Unity MR-Linac technology and further technical development of the MR-Linac system with the ultimate purpose to improve patients' survival, local, and regional tumor control and quality of life.

DETAILED DESCRIPTION:
Rationale: Radiation therapy has become indispensable in cancer treatment. However, it is associated with severe side effects. Innovation in radiation therapy has resulted in the development of MR-guided radiation therapy (MRGRT) which allows high precision radiotherapy under real time MR visualization. High precision MRGRT has the potential of dose escalation and margin reduction and may potentially lead to higher cure rates and less toxicity. MRGRT can be delivered by the MRI guided Linear Accelerator (MR-Linac) which integrates a state-of-the-art linear accelerator, 1.5T diagnostic quality MRI and an online adaptive workflow.

Objective: The Multi-OutcoMe EvaluatioN of radiation Therapy Using the MR-Linac Study (MOMENTUM) aims to accelerate the technical and clinical development of Anatomic and Biologic MRGRT and facilitate the evidence-based introduction of the MR-Linac into clinical practice. In MOMENTUM, technical and clinical data are gathered in order to optimize software, evaluate treatment outcomes, toxicities and progression free, disease free, and overall survival per disease site, and create a repository of anatomical and biological MR sequences to develop new features.

Study design: A multi-institutional, international observational cohort study. Study population: Cancer patients ≥ 18 years receiving treatment and/or imaging on an MR-Linac machine are eligible for enrollment.

Main study parameters/endpoints: MOMENTUM will collect technical and clinical patient data. The technical patient data is defined as data generated by (the use of) the MR-Linac and will include data collection during scans performed during routine care as well as research MRIs. Clinical data will be categorized into six classes: demographic, disease characteristics, treatment classifiers, toxicity outcomes, cancer control outcomes and PROs.

ELIGIBILITY:
Inclusion Criteria:

* Patient is to undergo or has completed imaging or treatment procedures on an MR-Linac;
* Patient provides written, informed consent;
* Patient is 18 years old or older.

Exclusion Criteria:

* MRI exclusion criteria, including
* MRI contraindications as per usual clinical care, such as (possible) pregnancy; claustrophobia and metal or electronic implants not compatible with MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment and/or imaging on an MR-Linac machine are eligible for enrolment. Patients must meet eligibility criteria and provide informed consent to be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | 3 months after MR-Linac treatment
  Progression free survival of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Progression-free Survival | 6 months after MR-Linac treatment
  Progression free survival of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Progression-free Survival | 24 months after MR-Linac treatment
  Progression free survival of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Survival | 3 months after MR-Linac treatment
  Overall survival of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Survival | 6 months after MR-Linac treatment
  Overall survival of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Survival | 24 months after MR-Linac treatment
  Overall survival of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Disease-free Survival | 3 months after MR-Linac treatment
  Disease-free survival of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Disease-free Survival | 6 months after MR-Linac treatment
  Disease-free survival of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Disease-free Survival | 24 months after MR-Linac treatment
  Disease-free survival of participating patients will be obtained from the hospital information systems. Patient follow-up is conducted to local standard of care practices.
Patient reported Health related quality of life (HRQoL). | 3 months after treatment.
  Patient reported health related quality of life is captured through a questionnaire the Generic European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30. They include 5 functional scales (physical, role, emotional, cognitive and social), three symptom scales, a global health scale, and six single items. All of these scales and items measures range in score from 0 to 100. A high score on functional or global health status scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Patient reported Health related quality of life (HRQoL). | 6 months after treatment.
  Patient reported health related quality of life is captured through a questionnaire the Generic European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30. They include 5 functional scales (physical, role, emotional, cognitive, and social), three symptom scales, a global health scale, and six single items. All of these scales and items measures range in score from 0 to 100. A high score on functional or global health status scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Patient reported Health related quality of life (HRQoL). | 12 months after treatment.
  Patient reported health related quality of life is captured through a questionnaire the Generic European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30. They include 5 functional scales (physical, role, emotional, cognitive and social), three symptom scales, a global health scale, and six single items. All of these scales and items measures range in score from 0 to 100. A high score on functional or global health status scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Patient reported Health related quality of life (HRQoL). | 24 months after treatment.
  Patient reported health related quality of life is captured through a questionnaire the Generic European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30. They include 5 functional scales (physical, role, emotional, cognitive and social), three symptom scales, a global health scale, and six single items. All of these scales and items measures range in score from 0 to 100. A high score on functional or global health status scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Patient reported Health related quality of life (HRQoL). | 3 months after treatment.
  Generic patient reported quality of life is captured by The EuroQol (EQ)-5D-5L questionnaire. This includes a descriptive system questionnaire and visual analogue scale (VAS). The descriptive system scores five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) from 1 to 5 where 1 means having no problems, and 5 means extreme problems or unable to participate. The digits can be combined in a 5-digit code to describe the overall health status. For example, 12111. The VAS records the overall current health on a vertical visual analogue scale from 0 to 100, respectively 'the worst health you can imagine' to 'the best health you can imagine'.
Patient reported Health related quality of life (HRQoL). | 6 months after treatment.
  Generic patient reported quality of life is captured by The EuroQol (EQ)-5D-5L questionnaire. This includes a descriptive system questionnaire and visual analogue scale (VAS). The descriptive system scores five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) from 1 to 5 where 1 means having no problems, and 5 means extreme problems or unable to participate. The digits can be combined in a 5-digit code to describe the overall health status. For example, 12111. The VAS records the overall current health on a vertical visual analogue scale from 0 to 100, respectively 'the worst health you can imagine' to 'the best health you can imagine'.
Patient reported Health related quality of life (HRQoL). | 12 months after treatment.
  Generic patient reported quality of life is captured by The EuroQol (EQ)-5D-5L questionnaire. This includes a descriptive system questionnaire and visual analogue scale (VAS). The descriptive system scores five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) from 1 to 5 where 1 means having no problems, and 5 means extreme problems or unable to participate. The digits can be combined in a 5-digit code to describe the overall health status. For example, 12111. The VAS records the overall current health on a vertical visual analogue scale from 0 to 100, respectively 'the worst health you can imagine' to 'the best health you can imagine'.
Patient reported Health related quality of life (HRQoL). | 24 months after treatment.
  Generic patient reported quality of life is captured by The EuroQol (EQ)-5D-5L questionnaire. This includes a descriptive system questionnaire and visual analogue scale (VAS). The descriptive system scores five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) from 1 to 5 where 1 means having no problems, and 5 means extreme problems or unable to participate. The digits can be combined in a 5-digit code to describe the overall health status. For example, 12111. The VAS records the overall current health on a vertical visual analogue scale from 0 to 100, respectively 'the worst health you can imagine' to 'the best health you can imagine'.
Patient reported tumor specific quality of life (QoL). | 3 months after treatment.
  Disease-specific patient reported quality of life is captured by a tumor specific EORTC QLQ questionnaire. (Brain-BN20, Breast-BR23, Bladder-BLM30, colorectal-CR29, Gynecological-CX24&VU34, Head and Neck-HN35, liver-HCC18 (primary) and -LMC21 (metastasis), lung-LC13, esophageal-OES18, prostate-PR2, pancreas-PAN26). They all include a different set of functional scales and symptom scales. All of these scales and items measures range in score from 0 to 100. A high score on functional scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Patient reported tumor specific quality of life (QoL). | 6 months after treatment.
  Disease-specific patient reported quality of life is captured by a tumor specific EORTC QLQ questionnaire. (Brain-BN20, Breast-BR23, Bladder-BLM30, colorectal-CR29, Gynecological-CX24&VU34, Head and Neck-HN35, liver-HCC18 (primary) and -LMC21 (metastasis), lung-LC13, esophageal-OES18, prostate-PR2, pancreas-PAN26). They all include a different set of functional scales and symptom scales. All of these scales and items measures range in score from 0 to 100. A high score on functional scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Patient reported tumor specific quality of life (QoL). | 12 months after treatment.
  Disease-specific patient reported quality of life is captured by a tumor specific EORTC QLQ questionnaire. (Brain-BN20, Breast-BR23, Bladder-BLM30, colorectal-CR29, Gynecological-CX24&VU34, Head and Neck-HN35, liver-HCC18 (primary) and -LMC21 (metastasis), lung-LC13, esophageal-OES18, prostate-PR2, pancreas-PAN26). They all include a different set of functional scales and symptom scales. All of these scales and items measures range in score from 0 to 100. A high score on functional scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Patient reported tumor specific quality of life (QoL). | 24 months after treatment.
  Disease-specific patient reported quality of life is captured by a tumor specific EORTC QLQ questionnaire. (Brain-BN20, Breast-BR23, Bladder-BLM30, colorectal-CR29, Gynecological-CX24&VU34, Head and Neck-HN35, liver-HCC18 (primary) and -LMC21 (metastasis), lung-LC13, esophageal-OES18, prostate-PR2, pancreas-PAN26). They all include a different set of functional scales and symptom scales. All of these scales and items measures range in score from 0 to 100. A high score on functional scale represents a high/healthy level of functioning. A high score for a symptom scale represents a high level of symptomatology.
Acute toxicity in common toxicity criteria for adverse events (CTCAE). | 3 months after treatment.
  Disease-specific toxicity is obtained from the hospital information system. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary.
Acute toxicity in common toxicity criteria for adverse events (CTCAE). | 6 months after treatment.
  Disease-specific toxicity is obtained from the hospital information system. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary.
Acute toxicity in common toxicity criteria for adverse events (CTCAE). | 12 months after treatment.
  Disease-specific toxicity is obtained from the hospital information system. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary.
Acute toxicity in common toxicity criteria for adverse events (CTCAE). | 24 months after treatment.
  Disease-specific toxicity is obtained from the hospital information system. Toxicities are reported according to the Common Terminology Criteria for Adverse Events (CTCAE) dictionary.
Clinical tumor response. | 2 year follow up.
  Clinical tumor response in participating patients is obtained from hospital information systems. Clinical patient follow-up and re-staging procedures are conducted to local standard of care practices.
Pathological tumor response. | 2 year follow up.
  Pathological tumor response in participating patients who undergo surgery are obtained from hospital information systems. Clinical patient follow-up and re-staging procedures are conducted to local standard of care practices.
Toxicity in common toxicity criteria for adverse events (CTCAE). | 2 years
  Disease-specific toxicity is obtained from the hospital information system.

CONTACTS AND LOCATIONS:
Overall Officials: Helena M Verkooijen, Prof, Dr, Principal Investigator — Universitair Medical Centre Utrecht
Locations (18):
- United States (3):
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - Md Anderson Cancer Center, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Austin Health - Olivia Newton-John Cancer Wellness and Research Centre, Melbourne, Australia
- Insitut Jules Bordet, Brussels, Belgium
- Canada (2):
  - Sunnybrook Health Sciences Centre/Odette Cancer Centre, Toronto, Ontario
  - University Health Network - Princess Margaret Cancer Center, Toronto
- Odense Universitetshospital, Odense, Funen, Denmark
- Universitätsklinikum Tübingen, Tübingen, Germany
- Italy (2):
  - Università degli Studi di Brescia, Brescia
  - IRCCS Ospedale Sacro Cuore Don Calabria, Negrar
- Netherlands (5):
  - Netherlands Cancer Institute, Antoni van Leeuwenhoek Hospital, Amsterdam
  - Radiotherapiegroep, Deventer
  - Radiotherapeutisch Instituut Friesland (RIF), Leeuwarden
  - Radboud UMC, Nijmegen
  - University Medical Center Utrecht, Utrecht
- United Kingdom (2):
  - The Royal Marsden and The Institute of Cancer Research National Institute for Health Research Biomedical Research Centre, London
  - The Christie National Health Service Foundation Trust, Manchester

REFERENCES:
- [Derived] Tan H, Stewart J, Ruschin M, Wang MH, Myrehaug S, Tseng CL, Detsky J, Husain Z, Chen H, Sahgal A, Soliman H. Inter-fraction dynamics during post-operative 5 fraction cavity hypofractionated stereotactic radiotherapy with a MR LINAC: a prospective serial imaging study. J Neurooncol. 2022 Feb;156(3):569-577. doi: 10.1007/s11060-021-03938-w. Epub 2022 Jan 3. PMID 34981300
- [Derived] de Mol van Otterloo SR, Christodouleas JP, Blezer ELA, Akhiat H, Brown K, Choudhury A, Eggert D, Erickson BA, Faivre-Finn C, Fuller CD, Goldwein J, Hafeez S, Hall E, Harrington KJ, van der Heide UA, Huddart RA, Intven MPW, Kirby AM, Lalondrelle S, McCann C, Minsky BD, Mook S, Nowee ME, Oelfke U, Orrling K, Sahgal A, Sarmiento JG, Schultz CJ, Tersteeg RJHA, Tijssen RHN, Tree AC, van Triest B, Hall WA, Verkooijen HM. The MOMENTUM Study: An International Registry for the Evidence-Based Introduction of MR-Guided Adaptive Therapy. Front Oncol. 2020 Sep 7;10:1328. doi: 10.3389/fonc.2020.01328. eCollection 2020. PMID 33014774